CLINICAL TRIAL: NCT06197789
Title: A Multi-center, Randomized, Independent Evaluator-Subject Blinded, Placebo-controlled, Phase 3 Clinical Study to Evaluate Safety and Efficacy of TPX-105 for Correction of Nasojugal Groove
Brief Title: Safety and Efficacy Study of TPX-105 for Correction of Nasojugal Groove
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tego Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-TPX-105-18-02
Record Dates: First submitted 2023-05-17; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Tear Trough Eyelid Deformity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPX-105 (Experimental): Autologous human dermal fibroblasts
  Interventions: Biological: TPX-105
- Placebo (Sham Comparator): Suspension media
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TPX-105 — Subjects will be administered with autologous fibroblasts through injection
  Other Names: Autologous human dermal fibroblasts
  Arms: TPX-105
Biological: Placebo — Subjects will be administered with Placebo through injection
  Arms: Placebo

SUMMARY:
Nasojugal groove correction is possible through surgical correction procedures, however, due to risks in safety and drawbacks not being able to be done on the young or after surgical procedure, dermal fillers which have the possibility of granulomatous allergic reaction and surface elevation. Therefore, there is a need for a safer procedure for nasojugal groove correction. This study evaluates the safety and efficacy of Autologous human dermal fibroblasts (TPX-105) used for the correction of nasojugal groove. The primary outcome is the improvement of nasojugal groove evaluated by an independent evaluator after administration of TPX-105 at week 24. Secondary outcomes include the improvement of nasojugal groove at week 4 and 12, severity change from baseline at week 4, 12 and 24 evaluated by an independent evaluator, and overall appearance improvement rate rated by subjects using Global Aesthetic Improvement Scale (GAIS) at week 4, 12, 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

Participants must;

1. Be 19 years old or older.
2. Have confirmed nasojugal groove severity equal to or more than "Moderate" (severity, grade 3) at subject assessment and want correction.
3. Consent to undergo skin biopsy on unexposed areas for manufacture of test product.
4. Fully understand the study and voluntarily sign the informed consent for participation in the study.

Exclusion Criteria:

Participants with any of the following conditions will be excluded unless stated otherwise;

1. Unsuitable for skin biopsy.

2. Have prior medical history of the following at the time of screening.

1. Keloids
2. Chronic skin diseases (psoriasis, atopic dermatis)
3. Genetic disorders that affect fibroblasts or collagen (ex. achondroplasia, osteogensis imperfecta, etc.)
4. Autoimmune disease
5. Human immunodeficiency virus (HIV) positive
6. Coagulopathy
7. Basal cell carcinoma or history of malignant tumors within the last 5 years

3. Have any of the following comorbidities at screening.

1. Inflammatory lesions or infectious diseases in the nasojugal groove region
2. Wounds, scars, or skin disorders that may affect efficacy assessment
3. Subjects who require continuous administration (2 weeks or more) of corticosteroid
4. Acute chronic infectious diseases
5. Subjects with bleeding requiring medical intervention including blood transfusions

4. Subjects who have a medical history of the following at the time of screening.

1. Surgical procedures or surgeries such as fillers or fat grafting on nasojugal groove or tear through deformity.
2. Surgical procedures or wrinkle corrections around the eyes within 24 weeks from screening. (Ex. botulinum toxin injection, face lift surgery, soft tissue augmentation, semi-intercalated peel, dermal photorejuvenation, or etc.)

5. Subjects who have received anti-platelet drugs and anticoagulants within 7 days prior to skin biopsy.

6. Subjects with planned facial cosmetic surgery (facial fillers, photorejuvenation, chemical/mechanical peeling) or facial massages during the duration of the study.

7. Subjects who have allergies to investigational drug composition or manufacturing ingredients (bovine proteins, gentamicin, etc.)

8. Be pregnant, breastfeeding, planning pregnancy or unwilling to use of contraceptive* suggested in this study.

*Hormonal contraceptives (oral, transplanted, etc.), intrauterine device, double-barrier method (condom, diaphragm, or cervical occlusive cap with spermicide), surgically sterile partner, etc.

9. Have participated in other clinical trials and received investigational agents within 4 weeks of this study.

10. Be deemed inadequate for the study by investigators. (Serious heart disease, liver disease, kidney disease, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Improvement Rate from Baseline | 24 weeks
  Improvement rate of nasojugal groove from baseline will be evaluated by a independent evaluator based on pictures taken at week 24 after administration of investigational product.
  *Improvement rate of nasojugal groove definition: With at least a 2-grade decrease

SECONDARY OUTCOMES:
Improvement Rate from Baseline | 4, 12 weeks
  Improvement rate of nasojugal groove from baseline evaluated by an independent evaluator based on pictures taken at week 4 and 12 after administration of investigational product.
Severity Grade Change from Baseline | 4, 12, 24 weeks
  Severity grade change from baseline evaluated by an independent evaluator based on pictures taken at week 4, 12 and 24 after administration of investigational product.
Overall Appearance Improvement Percentage (%) | 4, 12, 24, 48 weeks
  Overall appearance improvement percentage (%) rated by subjects using GAIS* at week 4, 12, 24 and 48 after administration of investigational product.
  *In the case of overall appearance improvement rate using GAIS being +2 points (Much Improved) or +1 (Improved)

CONTACTS AND LOCATIONS:
Overall Officials: Ho-yun Jun, Principal Investigator — Kyungpook National University Hospital
Locations (4):
- South Korea (4):
  - Soonchunhyang University Hospital Bucheon, Bucheon-si
  - Kyungpook National University Hospital, Daegu
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul